CLINICAL TRIAL: NCT00764205
Title: Randomized Trial of Prehospital Troponin Assessment Using the i-STAT Blood Analyzer
Brief Title: Randomized Trial of Prehospital Tropin Levels in Acute Coronary Syndrome (ACS)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Redmond Fire Department Medic One (Other Government)
Collaborators: Medic One Foundation (Other)
Responsible Party: James P. Jordan BS, MS, MICP, Redmond Fire Deparment Medic One
Other Study IDs: 20070224
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2008-10-01 (Estimated); Status verified 2008-09

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS; non STEMI; ECG troponin; iSTAT; Acute coronary syndrome without ST-segment elevation
MeSH Terms: conditions — Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study Group: Troponin measured prior to hospital arrival
- Control Group: Patients transported to hospital without troponin measurements enroute

SUMMARY:
This study randomizes patients seen by Redmond Medic One into a control arm and a study arm when they present with acute coronary syndrome and have non-contributory ECG's (i.e.non-STEMI). The control group is treated normally and delivered to the receiving hospital. The study group is treated normally as well, however troponin measurements are made using an i-STAT blood analyzer prior to hospital arrival. The results are presented to the receiving physician. Door-to-reperfusion time is monitored for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Over years of age
* ACS without ST-segment elevation
* Patient being transported to one of two participating hospitals

Exclusion Criteria:

* Less then 18 years of age.
* Post cardiac arrest.
* ACS with ST-segment elevation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen and treated by Redmond Fire Department Medic One.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Decrease door-to-reperfusion time for patients with non-STEMI's by measuring troponin levels prior to hospital arrival | 3-4 years

CONTACTS AND LOCATIONS:
Overall Officials: James P Jordan, BS, MS, MICP, Principal Investigator — Redmond Fire Department Medic One
Locations (1):
- Redmond Fire Department Medic One Units, -Mobile Units in King County-, Washington, United States